CLINICAL TRIAL: NCT01172899
Title: The BASIC Trial. Morbid Obesity in Children and Adolescents: a Prospective Randomised Trial of Conservative Treatment Versus Surgery
Brief Title: Bariatric Surgery in Children.
Acronym: BASIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL26279.068.09
Record Dates: First submitted 2010-07-22; First posted 2010-07-30 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Obesity, Morbid
Keywords: Bariatric Surgery; Adolescent
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic adjustable gastric band (Experimental)
  Interventions: Procedure: laparoscopic adjustable gastric band; Behavioral: Combined life style interventions
- Control group (Active Comparator)
  Interventions: Behavioral: Combined life style interventions

INTERVENTIONS:
Procedure: laparoscopic adjustable gastric band — Laparoscopic gastric band placement. Combined lifestyle interventions will continue after surgery.
  Arms: Laparoscopic adjustable gastric band
Behavioral: Combined life style interventions — Control group will receive standard therapy consisting of combined lifestyle interventions.

SUMMARY:
Rationale:

In the Western world overweight and obesity is an increasing problem both in adults and in children. In youth, it is associated with early death and a number of co-morbidities including metabolic and endocrine changes, increased inflammatory status, cardiovascular abnormalities, nonalcoholic fatty liver disease, and impaired quality of life.

The standard treatment for morbid obesity in children is by combined life style interventions. However, the medium and long term effects of dietetic interventions, behaviour therapy and medication is relatively poor. In adults bariatric surgery shows good results with up to 30% weight reduction in 3 years. The preliminary results in youth are similar, but surgery in this age group is relatively uncommon. In the Netherlands surgery in this age group is only allowed in clinical trials, until the benefits and risks have been established. (National Health Authorities)

Objective:

To determine if surgery gives a superior weight and body mass index (BMI) reduction than combined life style interventions in adolescents with morbid obesity and to assess its effect on obesity associated co-morbidity.

Study design:

Prospective randomised interventional study.

Study population:

Morbidly obese children, aged 14 - 16 years, with sex and age adjusted BMI >40 kg/m2 or >35 kg/m2 with co-morbidity.

Intervention:

Bariatric surgery by laparoscopic adjustable gastric band (LAGB) or combined life style interventions

Main study parameters/endpoints:

Primary endpoints: weight loss, loss of excess weight, loss of excess BMI. Secondary endpoints: Body composition, pubertal development, metabolic and endocrine changes, inflammatory status, cardiovascular abnormalities, non-alcoholic steatohepatitis, brain development, quality of life, and behaviour changes. The potential complications of surgery are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 to 16
* Age and sex adjusted BMI >40 kg/m2 or >35 kg/m2 with associated co-morbidity.

  * Associated co-morbidity includes: glucose intolerance, type 2 diabetes, hypertension, pseudotumor cerebri, acanthosis nigricans, obstructive sleep apnoea syndrome, depression, arthropathies, non-alcoholic steatohepatitis and dyslipidemia.
* > 1 year multidisciplinary organized weight reducing attempts with less than 5% weight loss
* Demonstrate decisional capacity

Exclusion Criteria:

* Psychologically not suitable
* Pre-menarche or bone age <15 years in boys
* Obesity associated to other disorders such as hypothyroidism
* Syndromal disorders such as Prader-Willi syndrome
* Severe cardiorespiratory impairment (ASA class 3 or higher)
* Insufficiently fluid in the Dutch language
* Unwillingness to adhere to follow-up programmes

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Weight | 6 months
  Weight loss, excess weight loss and loss of excess BMI.
Weight | 12 months
  Weight loss, excess weight loss and loss of excess BMI.
Weight | 24 months
  Weight loss, excess weight loss and loss of excess BMI.
Weight | 36 months
  Weight loss, excess weight loss and loss of excess BMI.

SECONDARY OUTCOMES:
Body composition | 12 months
  Next to anthropometric measurements, bone mineral content, bone density, lean bodymass and fat percentage will be assessed.
Pubertal development | 6 months
  Follow-up of hormonal status and Tanner stages.
Metabolic and endocrine changes | 6 months
Inflammatory status | 6 months
  Measurement of serum inflammatory markers.
Cardiovascular abnormalities | 6 months
Non-alcoholic fatty liver disease | 6 months
  Next to an ultrasound of the liver, serum levels of ALT, AST, ALP and GGT are measured. CCL-2 is used as a surrogate marker to assess liver disease.
Quality of life changes | 6 months
Behaviour changes | 6 months
  Measuring impulsivity and positive reward dominance with a computer task.
Operative complications | up to 36 months
  Early and late complications are being monitored
Effects on sleep architecture | 6 months
Brain development | 6 months
  If extra sponsorship can be gained, we will use fMRI and MEG in a subgroup to measure blood oxygen level-dependent (BOLD) brain response to food stimuli.
Body composition | 24 months
  Next to anthropometric measurements, bone mineral content, bone density, lean bodymass and fat percentage will be assessed.
Body composition | 36 months
  Next to anthropometric measurements, bone mineral content, bone density, lean bodymass and fat percentage will be assessed.
Pubertal development | 12 months
  Follow-up of hormonal status and Tanner stages.
Pubertal development | 24 months
  Follow-up of hormonal status and Tanner stages.
Pubertal development | 36 months
  Follow-up of hormonal status and Tanner stages.
Metabolic and endocrine changes | 12 months
Metabolic and endocrine changes | 24 months
Metabolic and endocrine changes | 36 months
Inflammatory status | 12 months
  Measurement of serum inflammatory markers.
Inflammatory status | 24 months
  Measurement of serum inflammatory markers.
Inflammatory status | 36 months
  Measurement of serum inflammatory markers.
Cardiovascular abnormalities | 12 months
Cardiovascular abnormalities | 24 months
Cardiovascular abnormalities | 36 months
Non-alcoholic fatty liver disease | 12 months
  Next to an ultrasound of the liver, serum levels of ALT, AST, ALP and GGT are measured. CCL-2 is used as a surrogate marker to assess liver disease.
Non-alcoholic fatty liver disease | 24 months
  Next to an ultrasound of the liver, serum levels of ALT, AST, ALP and GGT are measured. CCL-2 is used as a surrogate marker to assess liver disease.
Non-alcoholic fatty liver disease | 36 months
  Next to an ultrasound of the liver, serum levels of ALT, AST, ALP and GGT are measured. CCL-2 is used as a surrogate marker to assess liver disease.
Quality of life changes | 12 months
Quality of life changes | 24 months
Quality of life changes | 36 months
Effects on sleep architecture | 12 months
Effects on sleep architecture | 24 months
Effects on sleep architecture | 36 months
Behaviour changes | 12 months
  Measuring impulsivity and positive reward dominance with a computer task.
Behaviour changes | 24 months
  Measuring impulsivity and positive reward dominance with a computer task.
Behaviour changes | 36 months
  Measuring impulsivity and positive reward dominance with a computer task.
Brain development | 12 months
  If extra sponsorship can be gained, we will use fMRI and MEG in a subgroup to measure blood oxygen level-dependent (BOLD) brain response to food stimuli.
Brain development | 24 months
  If extra sponsorship can be gained, we will use fMRI and MEG in a subgroup to measure blood oxygen level-dependent (BOLD) brain response to food stimuli.
Brain development | 36 months
  If extra sponsorship can be gained, we will use fMRI and MEG in a subgroup to measure blood oxygen level-dependent (BOLD) brain response to food stimuli.
Physical activity | 6 months
  Assessment of physical activity using a questionnaire and an accelerometer.
Physical activity | 12 months
  Assessment of physical activity using a questionnaire and an accelerometer.
Physical activity | 24
  Assessment of physical activity using a questionnaire and an accelerometer.
Physical activity | 36 months
  Assessment of physical activity using a questionnaire and an accelerometer.
Behavior towards food | 6 months
  Behavior towards food is assessed by questionnaires and a computerized model for wanting and liking of food.
Behavior towards food | 12 months
  Behavior towards food is assessed by questionnaires and a computerized model for wanting and liking of food.
Behavior towards food | 24 months
  Behavior towards food is assessed by questionnaires and a computerized model for wanting and liking of food.
Behavior towards food | 36 months
  Behavior towards food is assessed by questionnaires and a computerized model for wanting and liking of food.

CONTACTS AND LOCATIONS:
Overall Officials: LWE van Heurn, Professor, Principal Investigator — Maastricht University Medical Center; Yvonne Roebroek, PhD Student, Principal Investigator — Maastricht University Medical Center; Givan F Paulus, PhD Student, Principal Investigator — Spaarne Gasthuis, Haarlem
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Roebroek YGM, Paulus GF, Talib A, van Mil EGAH, Vreugdenhil ACE, Winkens B, Stehouwer CDA, Greve JM, Bouvy ND, van Heurn LWE. Weight Loss and Glycemic Control After Bariatric Surgery in Adolescents With Severe Obesity: A Randomized Controlled Trial. J Adolesc Health. 2024 Mar;74(3):597-604. doi: 10.1016/j.jadohealth.2023.10.024. Epub 2023 Dec 9. PMID 38069930
- [Derived] Roebroek YGM, Paulus GF, van Mil EGAH, Vreugdenhil ACE, Winkens B, Nederkoorn C, Stehouwer CDA, Greve JWM, Bouvy ND, van Heurn LWE. Bariatric surgery in adolescents: a prospective randomized controlled trial comparing laparoscopic gastric banding to combined lifestyle interventions in adolescents with severe obesity (BASIC trial). BMC Pediatr. 2019 Jan 28;19(1):34. doi: 10.1186/s12887-019-1395-9. PMID 30691442
- See also: Study website (currently available in Dutch only) — http://www.basictrial.com